CLINICAL TRIAL: NCT00574548
Title: A Phase 3, Randomized, Active-Controlled, Modified Double-blind Trial to Evaluate the Safety, Tolerability, and Immunogenicity of 13-valent Pneumococcal Conjugate Vaccine When Administered Over 12 Months Either as a 2-Dose Regimen or With 23-valent Pneumococcal Polysaccharide Vaccine in Healthy Adults 60 to 64 Years of Age Who Are Naive to 23vPS
Brief Title: Study Evaluating the Safety, Tolerability and Immunogenicity of 13vPnC as a 2-Dose Regimen or With 23vPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 6115A1-3010; B1851027
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Pneumococcal Vaccines
Keywords: Vaccines, Pneumococcal Conjugate Vaccine
MeSH Terms: interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1.1 (Experimental): Group 1.1 = 13vPnC then 13vPnC
  Interventions: Biological: 13 valent Pneumococcal Conjugate Vaccine
- Group 1.2 (Experimental): Group 1.2 = 13vPnC then 23vPS
  Interventions: Biological: 13 valent Pneumococcal Conjugate Vaccine; Biological: 23-valent Pneumococcal Polysaccharide Vaccine
- Group 2 (Experimental): Group 2 = 23vPS then 13vPnC
  Interventions: Biological: 13 valent Pneumococcal Conjugate Vaccine; Biological: 23-valent Pneumococcal Polysaccharide Vaccine

INTERVENTIONS:
Biological: 13 valent Pneumococcal Conjugate Vaccine — 0.5 ml dose 13vPnC will be administered into the deltoid muscle at year 0 and year 1
  Arms: Group 1.1
Biological: 13 valent Pneumococcal Conjugate Vaccine — 0.5 ml dose 13vPnC will be administered into the deltoid muscle at year 0 and 0.5 ml dose 23vPS at year 1
  Arms: Group 1.2
Biological: 13 valent Pneumococcal Conjugate Vaccine — 0.5 ml dose 23vPS will be administered into the deltoid muscle at year 0 and 0.5 ml dose 13vPnC at year 1
  Arms: Group 2
Biological: 23-valent Pneumococcal Polysaccharide Vaccine — 0.5 ml dose 23vPS will be administered into the deltoid muscle at year 0 and 0.5 ml dose 13vPnC at year 1
  Arms: Group 2
Biological: 23-valent Pneumococcal Polysaccharide Vaccine — 0.5 ml dose 13vPnC will be administered into the deltoid muscle at year 0 and 0.5 ml dose 23vPS at year 1
  Arms: Group 1.2

SUMMARY:
The objective of this study is to compare the safety, tolerability and immunologic response to a dose of 23vPS or 13vPnC given one year after either 13vPnC or 23vPS in subjects that have never received a previous dose of 23vPS.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 60 to 64 years.
* Healthy.

Exclusion Criteria:

* Previous vaccination with any licensed or experimental pneumococcal vaccine.
* History of severe adverse reaction associated with a vaccine.
* Immunodeficiency.

Ages: 60 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 720 (Actual)
Dates: Start 2007-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Bristol, Tennessee

REFERENCES:
- [Derived] Greenberg RN, Gurtman A, Frenck RW, Strout C, Jansen KU, Trammel J, Scott DA, Emini EA, Gruber WC, Schmoele-Thoma B. Sequential administration of 13-valent pneumococcal conjugate vaccine and 23-valent pneumococcal polysaccharide vaccine in pneumococcal vaccine-naive adults 60-64 years of age. Vaccine. 2014 Apr 25;32(20):2364-74. doi: 10.1016/j.vaccine.2014.02.002. Epub 2014 Mar 5. PMID 24606865
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6115A1-3010&StudyName=Study%20Evaluating%20the%20Safety%2C%20Tolerability%20and%20Immunogenicity%20of%2013vPnC%20as%20a%202-Dose%20Regimen%20or%20with%2023vPS

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC - Group 1.1 or 1.2: Group 1.1: 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a single dose 0.5 milliliter (mL) intramuscularly (IM) at Year 0. 13vPnC administered as a single dose 0.5 mL IM at Year 1; or Group 1.2: 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a single dose 0.5 milliliter (mL) intramuscularly (IM) at Year 0. 23-valent polysaccharide vaccine (23vPS) administered as a single dose 0.5 mL IM at Year 1.
- 23vPS - Group 2: Group 2: 23vPS administered as a single dose 0.5 mL IM at Year 0. 13vPnC administered as a single dose 0.5 mL IM at Year 1.
Period: Overall Study
Arm/Group | 13vPnC - Group 1.1 or 1.2 | 23vPS - Group 2
Started | 482 | 238
Received Vaccination 1 (Vax 1) | 478 | 237
Completed Vax 1 (6 Month Contact) | 468 | 234
Withdrawn After Vax 1 (6 Month Contact) | 7 | 3
Withdrawn Before Vax 2 | 41 | 11
Received Vax 2 | 427 | 223
Completed Vax 2 (6 Month Contact) | 421 | 222
Completed | 421 | 222
Not Completed | 61 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC - Group 1.1 or 1.2 | 23vPS - Group 2 | Total
Number analyzed (Participants) | 478 | 237 | 715
Age Continuous [Mean (Standard Deviation); unit: years] | 61.7 (1.4) | 61.7 (1.4) | 61.7 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 281 | 134 | 415
  Male | 197 | 103 | 300

OUTCOME MEASURES:

1. Primary Outcome: Pneumococcal OPA Geometric Mean Titers (GMTs) for the 12 Common Serotypes for 13vPnC / 23vPS (Year 1) Versus 23vPS (Year 0)
Description: Antibody geometric mean titers as measured by opsonophagocytic assays (OPA) for 12 common pneumococcal serotypes (serotypes 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F). Confidence intervals (CI) for the GMTs are back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: 1 month after vaccination 1 (Vax 1=Day 1/ Year 0 [Visit 1]) and 1 month after vaccination 2 (Vax 2=Day 351 up to Day 379 after Visit 1)
Population: Evaluable immunogenicity population: participants who were eligible for the study, adhered to protocol requirements, had valid and determinate assay results, and had no major protocol violations. GMTs were calculated using all participants with available data for the specified blood draw.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Groups:
- 13vPnC / 23vPS: 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a single dose 0.5 milliliter (mL) intramuscularly (IM) at Year 0. 23-valent polysaccharide vaccine (23vPS) administered as a single dose 0.5 mL IM at Year 1.
- 23vPS: 23vPS administered as a single dose 0.5 mL IM at Year 0.
Arm/Group | 13vPnC / 23vPS | 23vPS
Number analyzed (Participants) | 233 | 229
geometric mean titer
  Common Serotype 1 | 148 [123.7 to 176.5] | 148 [117.9 to 185.9]
  Common Serotype 3 | 125 [108.6 to 143.4] | 80 [67.5 to 95.7]
  Common Serotype 4 | 1385 [1171.2 to 1638.7] | 1357 [1023.0 to 1799.0]
  Common Serotype 5 | 199 [161.4 to 246.2] | 140 [107.0 to 183.5]
  Common Serotype 6B | 1215 [965.4 to 1528.3] | 706 [522.1 to 954.0]
  Common Serotype 7F | 537 [422.4 to 682.6] | 331 [233.5 to 469.1]
  Common Serotype 9V | 373 [268.4 to 517.6] | 288 [198.0 to 419.1]
  Common Serotype 14 | 622 [485.7 to 796.4] | 734 [543.6 to 990.1]
  Common Serotype 18C | 1062 [863.2 to 1307.6] | 789 [586.2 to 1062.2]
  Common Serotype 19A | 467 [403.5 to 541.0] | 376 [302.8 to 465.7]
  Common Serotype 19F | 774 [642.0 to 933.6] | 509 [385.5 to 672.9]
  Common Serotype 23F | 198 [151.2 to 259.4] | 70 [49.9 to 97.3]
Statistical Analysis 1: Comparison: 13vPnC / 23vPS vs 23vPS; Serotype 1: ratio for GMT calculated by back transformation of the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — Criterion on which to declare non-inferiority = lower bound of the 2-sided 95% confidence interval for the geometric mean ratio greater than 0.5 (2-fold criterion); ratio of geometric mean titer = 1.0, 95% CI 2-sided [0.75 to 1.33] — CIs for the ratio are back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures ([13vPnC / 23vPS] - [23vPS])
Statistical Analysis 2: Comparison: 13vPnC / 23vPS vs 23vPS; Serotype 3: ratio for GMT calculated by back transformation of the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.6, 95% CI 2-sided [1.24 to 1.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC / 23vPS vs 23vPS; Serotype 4: ratio for GMT calculated by back transformation of the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.0, 95% CI 2-sided [0.74 to 1.41] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC / 23vPS vs 23vPS; Serotype 5: ratio for GMT calculated by back transformation of the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.4, 95% CI 2-sided [1.01 to 2.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC / 23vPS vs 23vPS; Serotype 6B: ratio for GMT calculated by back transformation of the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.7, 95% CI 2-sided [1.18 to 2.51] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC / 23vPS vs 23vPS; Serotype 7F: ratio for GMT calculated by back transformation of the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.6, 95% CI 2-sided [1.07 to 2.47] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC / 23vPS vs 23vPS; Serotype 9V: ratio for GMT calculated by back transformation of the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.3, 95% CI 2-sided [0.79 to 2.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC / 23vPS vs 23vPS; Serotype 14: ratio for GMT calculated by back transformation of the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 0.8, 95% CI 2-sided [0.58 to 1.25] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC / 23vPS vs 23vPS; Serotype 18C: ratio for GMT calculated by back transformation of the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.3, 95% CI 2-sided [0.94 to 1.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC / 23vPS vs 23vPS; Serotype 19A: ratio for GMT calculated by back transformation of the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.2, 95% CI 2-sided [0.96 to 1.61] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC / 23vPS vs 23vPS; Serotype 19F: ratio for GMT calculated by back transformation of the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.5, 95% CI 2-sided [1.09 to 2.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC / 23vPS vs 23vPS; Serotype 23F: ratio for GMT calculated by back transformation of the mean difference between vaccine groups on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 2.8, 95% CI 2-sided [1.86 to 4.35] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Pneumococcal OPA Geometric Mean Titers (GMTs) for the 12 Common Serotypes for 13vPnC / 23vPS Versus 23vPS / 13vPnC (Year 1)
Description: as for outcome 1
Time Frame: 1 month after vaccination 2 (Vax 2=Day 351 up to Day 379 after Visit 1)
Population: Evaluable immunogenicity population. GMTs were calculated using all participants with available data for the specified blood draw.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Groups:
- 23vPS / 13vPnC: 23vPS administered as a single dose 0.5 mL IM at Year 0. 13vPnC administered as a single dose 0.5 mL IM at Year 1.
Arm/Group | 13vPnC / 23vPS | 23vPS / 13vPnC
Number analyzed (Participants) | 233 | 196
geometric mean titer
  Common Serotype 1 | 148 [123.7 to 176.5] | 77 [60.7 to 98.1]
  Common Serotype 3 | 125 [108.6 to 143.4] | 50 [40.9 to 61.7]
  Common Serotype 4 | 1385 [1171.2 to 1638.7] | 935 [739.9 to 1182.4]
  Common Serotype 5 | 199 [161.4 to 246.2] | 85 [64.2 to 112.0]
  Common Serotype 6B | 1215 [965.4 to 1528.3] | 710 [529.1 to 953.2]
  Common Serotype 7F | 537 [422.4 to 682.6] | 126 [85.6 to 184.6]
  Common Serotype 9V | 373 [268.4 to 517.6] | 114 [76.5 to 169.3]
  Common Serotype 14 | 622 [485.7 to 796.4] | 435 [323.0 to 585.7]
  Common Serotype 18C | 1062 [863.2 to 1307.6] | 564 [418.2 to 761.7]
  Common Serotype 19A | 467 [403.5 to 541.0] | 289 [235.7 to 353.9]
  Common Serotype 19F | 774 [642.0 to 933.6] | 286 [217.3 to 376.7]
  Common Serotype 23F | 198 [151.2 to 259.4] | 124 [88.2 to 173.0]
Statistical Analysis 1: Comparison: 13vPnC / 23vPS vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.9, 95% CI 2-sided [1.43 to 2.57] — CIs for the ratio are back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures ([13vPnC / 23vPS] - [23vPS / 13vPnC])
Statistical Analysis 2: Comparison: 13vPnC / 23vPS vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 2.5, 95% CI 2-sided [1.95 to 3.16] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC / 23vPS vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.5, 95% CI 2-sided [1.12 to 1.96] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC / 23vPS vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 2.4, 95% CI 2-sided [1.67 to 3.31] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC / 23vPS vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.7, 95% CI 2-sided [1.19 to 2.47] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC / 23vPS vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 6]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 4.3, 95% CI 2-sided [2.76 to 6.61] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC / 23vPS vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 7]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 3.3, 95% CI 2-sided [1.97 to 5.45] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC / 23vPS vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.4, 95% CI 2-sided [0.98 to 2.10] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC / 23vPS vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.9, 95% CI 2-sided [1.32 to 2.69] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC / 23vPS vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 10]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.6, 95% CI 2-sided [1.27 to 2.07] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC / 23vPS vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 11]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 2.7, 95% CI 2-sided [1.96 to 3.74] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC / 23vPS vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 12]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ratio of geometric mean titer = 1.6, 95% CI 2-sided [1.05 to 2.45] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Pneumococcal OPA Geometric Mean Titers (GMTs) for the 13 Serotypes for 13vPnC / 13vPnC (Year 1) Versus 13vPnC (Year 0)
Description: Antibody geometric mean titers as measured by opsonophagocytic assays (OPA) for the pneumococcal serotypes (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F). The 6A pneumococcal serotype is specific to 13vPnC. Confidence intervals (CI) for the GMTs are back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: as for outcome 1
Population: Evaluable immunogenicity population. GMTs were calculated using all participants with available data who had determinate assay values at both the postvaccination 1 (13vPnC; Year 0) and postvaccination 2 (13vPnC / 13vPnC; Year 1) time points.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Groups:
- 13vPnC Vaccination 1 (Year 0): 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a single dose 0.5 milliliter (mL) intramuscularly (IM) at Year 0.
- 13vPnC / 13vPnC Vaccination 2 (Year 1): 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a single dose 0.5 milliliter (mL) intramuscularly (IM) at Year 0. 13vPnC administered as a single dose 0.5 mL IM at Year 1.
Arm/Group | 13vPnC Vaccination 1 (Year 0) | 13vPnC / 13vPnC Vaccination 2 (Year 1)
Number analyzed (Participants) | 127 | 127
geometric mean titer
  Common Serotype 1 | 215 [163.9 to 282.4] | 142 [112.2 to 180.4]
  Common Serotype 3 | 73 [57.2 to 94.1] | 89 [75.2 to 105.4]
  Common Serotype 4 | 2255 [1625.2 to 3128.6] | 1214 [931.8 to 1582.1]
  Common Serotype 5 | 170 [112.1 to 258.6] | 98 [69.6 to 136.6]
  Additional Serotype 6A | 2682 [1969.5 to 3652.1] | 2281 [1747.1 to 2978.5]
  Common Serotype 6B | 2112 [1508.0 to 2958.2] | 1882 [1429.7 to 2477.9]
  Common Serotype 7F | 930 [602.1 to 1437.1] | 323 [215.8 to 482.8]
  Common Serotype 9V | 919 [619.1 to 1364.0] | 335 [214.6 to 522.6]
  Common Serotype 14 | 492 [312.7 to 774.5] | 384 [262.4 to 561.2]
  Common Serotype 18C | 1440 [1015.3 to 2043.5] | 986 [730.8 to 1330.2]
  Common Serotype 19A | 583 [426.6 to 796.8] | 385 [308.2 to 481.6]
  Common Serotype 19F | 566 [385.7 to 829.2] | 502 [381.3 to 662.1]
  Common Serotype 23F | 291 [187.7 to 452.2] | 456 [322.4 to 644.7]
Statistical Analysis 1: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 13vPnC Vaccination 2 (Year 1); Serotype 1: geometric mean fold rise (GMFR) calculated using all evaluable participants with data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — Criterion on which to declare non-inferiority = lower bound of the 2-sided 95% confidence interval for the geometric mean fold rise greater than 0.5; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.54 to 0.82] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 2: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 13vPnC Vaccination 2 (Year 1); Serotype 3: geometric mean fold rise (GMFR) calculated using all evaluable participants with data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 1.2, 95% CI 2-sided [0.99 to 1.49] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 3: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 13vPnC Vaccination 2 (Year 1); Serotype 4: geometric mean fold rise (GMFR) calculated using all evaluable participants with data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.43 to 0.68] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 4: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 13vPnC Vaccination 2 (Year 1); Serotype 5: geometric mean fold rise (GMFR) calculated using all evaluable participants with data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.43 to 0.77] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 5: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 13vPnC Vaccination 2 (Year 1); Serotype 6A: geometric mean fold rise (GMFR) calculated using all evaluable participants with data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.67 to 1.08] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 6: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 13vPnC Vaccination 2 (Year 1); Serotype 6B: geometric mean fold rise (GMFR) calculated using all evaluable participants with data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.71 to 1.12] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 7: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 13vPnC Vaccination 2 (Year 1); Serotype 7F: geometric mean fold rise (GMFR) calculated using all evaluable participants with data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.24 to 0.49] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 8: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 13vPnC Vaccination 2 (Year 1); Serotype 9V: geometric mean fold rise (GMFR) calculated using all evaluable participants with data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.26 to 0.51] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 9: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 13vPnC Vaccination 2 (Year 1); Serotype 14: geometric mean fold rise (GMFR) calculated using all evaluable participants with data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.8, 95% CI 2-sided [0.60 to 1.02] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 10: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 13vPnC Vaccination 2 (Year 1); Serotype 18C: geometric mean fold rise (GMFR) calculated using all evaluable participants with data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.54 to 0.87] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 11: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 13vPnC Vaccination 2 (Year 1); Serotype 19A: geometric mean fold rise (GMFR) calculated using all evaluable participants with data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.53 to 0.82] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 12: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 13vPnC Vaccination 2 (Year 1); Serotype 19F: geometric mean fold rise (GMFR) calculated using all evaluable participants with data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.69 to 1.15] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 13: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 13vPnC Vaccination 2 (Year 1); Serotype 23F: geometric mean fold rise (GMFR) calculated using all evaluable participants with data from both the postvaccination 1 and postvaccination 2 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 1.6, 95% CI 2-sided [1.15 to 2.13] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise

4. Secondary Outcome: Pneumococcal OPA Geometric Mean Titers (GMTs) for the 12 Common Serotypes for 13vPnC / 23vPS (Year 1) Versus 13vPnC (Year 0)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Evaluable immunogenicity population. GMTs were calculated using all participants with available data who had determinate assay values at both the postvaccination 1 (13vPnC; Year 0) and postvaccination 2 (13vPnC / 23vPS; Year 1) time points.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Groups:
- 13vPnC / 23vPS Vaccination 2 (Year 1): 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a single dose 0.5 milliliter (mL) intramuscularly (IM) at Year 0. 23-valent polysaccharide vaccine (23vPS) administered as a single dose 0.5 mL IM at Year 1.
Arm/Group | 13vPnC Vaccination 1 (Year 0) | 13vPnC / 23vPS Vaccination 2 (Year 1)
Number analyzed (Participants) | 221 | 221
geometric mean titer
  Common Serotype 1 | 220 [178.9 to 269.3] | 140 [117.4 to 168.1]
  Common Serotype 3 | 74 [61.3 to 88.7] | 129 [112.4 to 147.5]
  Common Serotype 4 | 2517 [2091.7 to 3029.2] | 1430 [1214.7 to 1683.9]
  Common Serotype 5 | 227 [170.9 to 300.5] | 188 [151.1 to 234.8]
  Common Serotype 6B | 2012 [1571.9 to 2574.1] | 1351 [1087.6 to 1677.0]
  Common Serotype 7F | 1252 [971.1 to 1614.4] | 533 [419.2 to 678.2]
  Common Serotype 9V | 758 [563.8 to 1018.9] | 406 [292.3 to 564.6]
  Common Serotype 14 | 664 [485.1 to 908.5] | 616 [473.3 to 802.2]
  Common Serotype 18C | 1532 [1183.7 to 1982.7] | 1074 [871.7 to 1322.2]
  Common Serotype 19A | 696 [581.1 to 833.6] | 457 [389.5 to 536.3]
  Common Serotype 19F | 696 [546.3 to 887.7] | 773 [636.6 to 937.6]
  Common Serotype 23F | 358 [265.5 to 481.7] | 216 [165.0 to 282.7]
Statistical Analysis 1: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 23vPS Vaccination 2 (Year 1); [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.55 to 0.75] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 2: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 23vPS Vaccination 2 (Year 1); [analysis description as in outcome 3, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 1.7, 95% CI 2-sided [1.52 to 2.01] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 3: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 23vPS Vaccination 2 (Year 1); [analysis description as in outcome 3, analysis 3]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.49 to 0.66] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 4: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 23vPS Vaccination 2 (Year 1); [analysis description as in outcome 3, analysis 4]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.8, 95% CI 2-sided [0.67 to 1.03] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 5: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 23vPS Vaccination 2 (Year 1); [analysis description as in outcome 3, analysis 6]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.57 to 0.79] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 6: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 23vPS Vaccination 2 (Year 1); [analysis description as in outcome 3, analysis 7]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.35 to 0.52] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 7: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 23vPS Vaccination 2 (Year 1); [analysis description as in outcome 3, analysis 8]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.41 to 0.69] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 8: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 23vPS Vaccination 2 (Year 1); [analysis description as in outcome 3, analysis 9]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.75 to 1.15] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 9: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 23vPS Vaccination 2 (Year 1); [analysis description as in outcome 3, analysis 10]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.58 to 0.85] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 10: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 23vPS Vaccination 2 (Year 1); [analysis description as in outcome 3, analysis 11]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.58 to 0.74] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 11: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 23vPS Vaccination 2 (Year 1); [analysis description as in outcome 3, analysis 12]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 1.1, 95% CI 2-sided [0.89 to 1.39] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 12: Comparison: 13vPnC Vaccination 1 (Year 0) vs 13vPnC / 23vPS Vaccination 2 (Year 1); [analysis description as in outcome 3, analysis 13]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.50 to 0.73] — CIs are back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise

5. Other Pre Specified Outcome: Pneumococcal OPA Geometric Mean Titers (GMTs) for the 12 Common Serotypes for 23vPS / 13vPnC (Year 1) Versus 13vPnC (Year 0)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Groups:
- 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a single dose 0.5 milliliter (mL) intramuscularly (IM) at Year 0.
Arm/Group | 13vPnC | 23vPS / 13vPnC
Number analyzed (Participants) | 455 | 196
geometric mean titer
  Common Serotype 1 | 207 [177.7 to 240.9] | 77 [60.7 to 98.1]
  Common Serotype 3 | 75 [66.0 to 85.3] | 50 [40.9 to 61.7]
  Common Serotype 4 | 2536 [2192.3 to 2933.0] | 935 [739.9 to 1182.4]
  Common Serotype 5 | 215 [175.9 to 261.7] | 85 [64.2 to 112.0]
  Common Serotype 6B | 1948 [1614.0 to 2351.7] | 710 [529.1 to 953.2]
  Common Serotype 7F | 1063 [868.6 to 1302.2] | 126 [85.6 to 184.6]
  Common Serotype 9V | 767 [620.0 to 949.3] | 114 [76.5 to 169.3]
  Common Serotype 14 | 650 [524.9 to 805.8] | 435 [323.0 to 585.7]
  Common Serotype 18C | 1576 [1321.3 to 1880.9] | 564 [418.2 to 761.7]
  Common Serotype 19A | 709 [618.9 to 811.2] | 289 [235.7 to 353.9]
  Common Serotype 19F | 711 [595.9 to 848.9] | 286 [217.3 to 376.7]
  Common Serotype 23F | 354 [283.8 to 440.7] | 124 [88.2 to 173.0]
Statistical Analysis 1: Comparison: 13vPnC vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ratio of geometric mean titer = 2.7, 95% CI 2-sided [2.03 to 3.55] — CIs for the ratio are back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures ([13vPnC] - [23vPS / 13vPnC])
Statistical Analysis 2: Comparison: 13vPnC vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; ratio of geometric mean titer = 1.5, 95% CI 2-sided [1.18 to 1.89] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; ratio of geometric mean titer = 2.7, 95% CI 2-sided [2.07 to 3.55] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; ratio of geometric mean titer = 2.5, 95% CI 2-sided [1.77 to 3.61] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; ratio of geometric mean titer = 2.7, 95% CI 2-sided [1.94 to 3.88] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; ratio of geometric mean titer = 8.5, 95% CI 2-sided [5.68 to 12.60] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; ratio of geometric mean titer = 6.7, 95% CI 2-sided [4.45 to 10.22] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; ratio of geometric mean titer = 1.5, 95% CI 2-sided [1.02 to 2.18] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; ratio of geometric mean titer = 2.8, 95% CI 2-sided [2.01 to 3.89] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; ratio of geometric mean titer = 2.5, 95% CI 2-sided [1.92 to 3.13] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; ratio of geometric mean titer = 2.5, 95% CI 2-sided [1.80 to 3.44] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC vs 23vPS / 13vPnC; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; ratio of geometric mean titer = 2.9, 95% CI 2-sided [1.92 to 4.28] — [estimate comment as in outcome 5, analysis 1]

6. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination 1 (Year 0) 13vPnC and 23vPS
Description: Local reactions reported using an electronic diary. Redness and Swelling scaled as Any (redness present or swelling present); Mild (2.5 to 5.0 centimeters [cm]; Moderate (5.1 to 10.0 cm); Severe (>10 cm). Pain scaled as Any (pain present); Mild (awareness of pain; easily tolerated); Moderate (discomfort enough to cause interference with usual activity); Severe (incapacitating); Limitation of arm movement scaled as Any (limitation present); Mild (some limitation); Moderate (unable to move arm above head; able to move arm above shoulder); Severe (unable to move arm above shoulder).
Time Frame: 14 days after vaccination 1 (Vax 1=Day 1/ Year 0 [Visit 1]) and 14 days after vaccination 2 (Vax 2=Day 351 up to Day 379 after Visit 1)
Population: Safety population includes all participants who receive at least 1 dose of study vaccine. N=number of participants with any local reaction; (n)=number of participants with known values for 13vPnC and 23vPS, respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 23vPS
Number analyzed (Participants) | 374 | 180
percentage of participants
  Redness: Any (n=270, 134) | 12.2 | 11.2
  Redness: Mild (n=266, 134) | 8.3 | 9.7
  Redness: Moderate (n=264, 128) | 6.4 | 3.9
  Redness: Severe (n=259, 127) | 1.2 | 0.8
  Swelling: Any (n=270, 135) | 10.0 | 10.4
  Swelling: Mild (n=268, 132) | 8.2 | 6.1
  Swelling: Moderate (n=263, 132) | 3.8 | 7.6
  Swelling: Severe (n=258, 127) | 0.0 | 0.0
  Pain: Any (n=370, 175) | 69.2 | 58.3
  Pain: Mild (n=360, 170) | 66.1 | 52.9
  Pain: Moderate (n=284, 143) | 20.1 | 21.7
  Pain: Severe (n=261, 127) | 2.3 | 0.8
  Limitation of arm movement: Any (n=289, 142) | 23.5 | 28.2
  Limitation of arm movement: Mild (n=286, 142) | 22.7 | 26.1
  Limitation of arm movement: Moderate (n=260, 127) | 1.2 | 3.1
  Limitation of arm movement: Severe (n=261, 128) | 1.1 | 2.3

7. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1)
Description: as for outcome 6
Time Frame: as for outcome 6
Population: Safety population; N=number of participants with any local reaction; (n)=number of participants with known values for 13vPnC and 13vPnC / 13vPnC, respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC / 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a single dose 0.5 milliliter (mL) intramuscularly (IM) at Year 0. 13vPnC administered as a single dose 0.5 mL IM at Year 1.
Arm/Group | 13vPnC | 13vPnC / 13vPnC
Number analyzed (Participants) | 110 | 110
percentage of participants
  Redness: Any (n=61, 61) | 14.8 | 11.5
  Redness: Mild (n=57, 57) | 7.0 | 8.8
  Redness: Moderate (n=58, 58) | 8.6 | 3.4
  Redness: Severe (n=57, 57) | 0.0 | 3.5
  Swelling: Any (n=60, 60) | 10.0 | 11.7
  Swelling: Mild (n=59, 59) | 6.8 | 8.5
  Swelling: Moderate (n=55, 55) | 1.8 | 3.6
  Swelling: Severe (n=56, 56) | 0.0 | 1.8
  Pain: Any (n=108, 108) | 76.9 | 75.9
  Pain: Mild (n=101, 101) | 72.3 | 72.3
  Pain: Moderate (n=61, 61) | 21.3 | 26.2
  Pain: Severe (n=57, 57) | 0.0 | 3.5
  Limitation of arm movement: Any (n=65, 65) | 26.2 | 24.6
  Limitation of arm movement: Mild (n=65, 65) | 26.2 | 24.6
  Limitation of arm movement: Moderate (n=56, 56) | 1.8 | 0.0
  Limitation of arm movement: Severe (n=56, 56) | 0.0 | 1.8

8. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1)
Description: as for outcome 6
Time Frame: as for outcome 6
Population: Safety population; N=number of participants with any local reaction; (n)=number of participants with known values for 13vPnC and 23vPS / 13vPnC, respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 23vPS / 13vPnC
Number analyzed (Participants) | 374 | 171
percentage of participants
  Redness: Any (n=270, 115) | 12.2 | 4.3
  Redness: Mild (n=266, 115) | 8.3 | 4.3
  Redness: Moderate (n=264, 115) | 6.4 | 0.9
  Redness: Severe (n=259, 115) | 1.2 | 0.0
  Swelling: Any (n=270, 119) | 10.0 | 5.0
  Swelling: Mild (n=268, 119) | 8.2 | 5.0
  Swelling: Moderate (n=263, 116) | 3.8 | 0.9
  Swelling: Severe (n=258, 115) | 0.0 | 0.0
  Pain: Any (n=370, 169) | 69.2 | 69.8
  Pain: Mild (n=360, 166) | 66.1 | 68.1
  Pain: Moderate (n=284, 129) | 20.1 | 17.8
  Pain: Severe (n=261, 116) | 2.3 | 0.9
  Limitation of arm movement: Any (n=289, 130) | 23.5 | 18.5
  Limitation of arm movement: Mild (n=286, 130) | 22.7 | 16.9
  Limitation of arm movement: Moderate (n=260, 115) | 1.2 | 0.0
  Limitation of arm movement: Severe (n=261, 115) | 1.1 | 1.7

9. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination 23vPS (Year 0) and 13vPnC / 23vPS (Year 1)
Description: Local reactions reported using an electronic diary. Redness and Swelling scaled as Any (redness present or swelling present); Mild (2.5 to 5.0 centimeters [cm]); Moderate (5.1 to 10.0 cm); Severe (>10 cm). Pain scaled as Any (pain present); Mild (awareness of pain; easily tolerated); Moderate (discomfort enough to cause interference with usual activity); Severe (incapacitating); Limitation of arm movement scaled as Any (limitation present); Mild (some limitation); Moderate (unable to move arm above head; able to move arm above shoulder); Severe (unable to move arm above shoulder).
Time Frame: as for outcome 6
Population: Safety population; N=number of participants with any local reaction; (n)=number of participants with known values for 23vPS and 13vPnC / 23vPS, respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 23vPS | 13vPnC / 23vPS
Number analyzed (Participants) | 180 | 234
percentage of participants
  Redness: Any (n=134, 151) | 11.2 | 27.8
  Redness: Mild (n=134, 144) | 9.7 | 19.4
  Redness: Moderate (n=128, 138) | 3.9 | 12.3
  Redness: Severe (n=127, 131) | 0.8 | 6.9
  Swelling: Any (n=135, 155) | 10.4 | 25.8
  Swelling: Mild (n=132, 149) | 6.1 | 20.1
  Swelling: Moderate (n=132, 138) | 7.6 | 12.3
  Swelling: Severe (n=127, 132) | 0.0 | 6.1
  Pain: Any (n=175, 231) | 58.3 | 85.7
  Pain: Mild (n=170, 205) | 52.9 | 78.5
  Pain: Moderate (n=143, 176) | 21.7 | 49.4
  Pain: Severe (n=127, 140) | 0.8 | 12.9
  Limitation of arm movement: Any (n=142, 178) | 28.2 | 53.4
  Limitation of arm movement: Mild (n=142, 171) | 26.1 | 47.4
  Limitation of arm movement: Moderate (n=127, 134) | 3.1 | 10.4
  Limitation of arm movement: Severe (n=128, 135) | 2.3 | 8.1

10. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination 2 (Year 1) 13vPnC / 13vPnC, 13vPnC / 23vPS, and 23vPS / 13vPnC
Description: as for outcome 6
Time Frame: 14 days after vaccination 2 (Vax 2=Day 351 up to Day 379 after Visit 1)
Population: Safety population; N=number of participants with any local reaction; (n)=number of participants with known values for 13vPnC / 13vPnC, 13vPnC / 23vPS, and 23vPS / 13vPnC, respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC / 13vPnC | 13vPnC / 23vPS | 23vPS / 13vPnC
Number analyzed (Participants) | 130 | 234 | 171
percentage of participants
  Redness: Any (n=86, 151, 115) | 12.8 | 27.8 | 4.3
  Redness: Mild (n=83, 144, 115) | 7.2 | 19.4 | 4.3
  Redness: Moderate (n=83, 138, 115) | 7.2 | 12.3 | 0.9
  Redness: Severe (n=83, 131, 115) | 2.4 | 6.9 | 0.0
  Swelling: Any (n=86, 155, 119) | 14.0 | 25.8 | 5.0
  Swelling: Mild (n=85, 149, 119) | 10.6 | 20.1 | 5.0
  Swelling: Moderate (n=82, 138, 116) | 6.1 | 12.3 | 0.9
  Swelling: Severe (n=82, 132, 115) | 1.2 | 6.1 | 0.0
  Pain: Any (n=129, 231, 169) | 75.2 | 85.7 | 69.8
  Pain: Mild (n=123, 205, 166) | 72.4 | 78.5 | 68.1
  Pain: Moderate (n=91, 176, 129) | 24.2 | 49.4 | 17.8
  Pain: Severe (n=83, 140, 116) | 2.4 | 12.9 | 0.9
  Limitation of arm movement: Any (n=93, 178, 130) | 28.0 | 53.4 | 18.5
  Limitation of arm movement: Mild (n=92, 171, 130) | 27.2 | 47.4 | 16.9
  Limitation of arm movement: Moderate(n=83,134,115) | 3.6 | 10.4 | 0.0
  Limitation of arm movement: Severe (n=82, 135,115) | 1.2 | 8.1 | 1.7

11. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination 1 (Year 0) 13vPnC and 23vPS
Description: Systemic events reported using an electronic diary. Systemic events are any fever ≥38 degrees Celsius [C], fatigue, headache, chills, rash, vomiting, decreased appetite, new generalized muscle pain (new muscle pain), aggravated generalized muscle pain (aggravated muscle pain), new generalized joint pain (new joint pain), and aggravated generalized joint pain (aggravated joint pain). Participants may be represented in more than 1 category.
Time Frame: 14 days after vaccination 1 (Vax 1=Day 1/ Year 0 [Visit 1])
Population: Safety population; N=number of participants with any systemic event; (n)=number of participants with known values for 13vPnC and 23vPS, respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 23vPS
Number analyzed (Participants) | 383 | 202
percentage of participants
  Fever: Any ≥38 degrees C (n=263, 127) | 4.6 | 1.6
  Fever: Mild ≥38 but <38.5 degrees C (n=263, 127) | 3.8 | 0.8
  Fever: Moderate ≥38.5 but <39 degrees C(n=259,127) | 0.8 | 0.0
  Fever: Severe ≥39 but ≤40 degrees C (n=259, 127) | 0.4 | 0.8
  Fever Potentially life threatening >40C(n=258,127) | 0.4 | 0.0
  Fatigue (n=321, 173) | 50.5 | 49.1
  Headache (n=328, 167) | 49.7 | 46.1
  Chills (n=286, 145) | 19.9 | 26.9
  Rash (n=267, 134) | 8.6 | 13.4
  Vomiting (n=261, 131) | 3.1 | 3.1
  Decreased appetite (n=278, 148) | 14.7 | 23.0
  New muscle pain (n=324, 167) | 46.9 | 51.5
  Aggravated muscle pain (n=286, 154) | 22.0 | 32.5
  New joint pain (n=278, 147) | 15.5 | 23.81
  Aggravated joint pain (n=272, 142) | 14.0 | 21.1

12. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1)
Description: as for outcome 11
Time Frame: as for outcome 6
Population: Safety population; N=number of participants with any systemic event; (n)=number of participants with known values for 13vPnC and 13vPnC / 13vPnC, respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 13vPnC / 13vPnC
Number analyzed (Participants) | 102 | 102
percentage of participants
  Fever: Any ≥38 degrees C (n=55, 55) | 9.1 | 3.6
  Fever: Mild ≥38 but <38.5 degrees C (n=55, 55) | 7.3 | 0.0
  Fever: Moderate ≥38.5 but <39 degrees C(n=55, 55) | 0.0 | 1.8
  Fever: Severe ≥39 but ≤40 degrees C (n=55, 55) | 0.0 | 0.0
  Fever Potentially life threatening >40C (n=55, 55) | 1.8 | 1.8
  Fatigue (n=76, 76) | 56.6 | 43.4
  Headache (n=76, 76) | 52.6 | 44.7
  Chills (n=61, 61) | 18.0 | 19.7
  Rash (n=60, 60) | 8.3 | 10.0
  Vomiting (n=56, 56) | 7.1 | 3.6
  Decreased appetite (n=61, 61) | 13.1 | 21.3
  New muscle pain (n=84, 84) | 47.6 | 51.2
  Aggravated muscle pain (n=68, 68) | 26.5 | 30.9
  New joint pain (n=62, 62) | 14.5 | 16.1
  Aggravated joint pain (n=62, 62) | 16.1 | 19.4

13. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1)
Description: as for outcome 11
Time Frame: as for outcome 6
Population: Safety population; N=number of participants with any systemic event; (n)=number of participants with known values for 13vPnC and 23vPS / 13vPnC , respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 23vPS / 13vPnC
Number analyzed (Participants) | 383 | 169
percentage of participants
  Fever: Any ≥38 degrees C (n=263, 116) | 4.6 | 0.9
  Fever: Mild ≥38 but <38.5 degrees C (n=263, 116) | 3.8 | 0.9
  Fever: Moderate ≥38.5 but <39 degrees C(n=259,115) | 0.8 | 0.0
  Fever: Severe ≥39 but ≤40 degrees C(n=259,115) | 0.4 | 0.0
  Fever Potentially life threatening >40C(n=258,115) | 0.4 | 0.0
  Fatigue (n=321, 141) | 50.5 | 41.1
  Headache (n=328, 139) | 49.7 | 40.3
  Chills (n=286, 127) | 19.9 | 19.7
  Rash (n=267, 121) | 8.6 | 8.3
  Vomiting (n=261, 118) | 3.1 | 6.8
  Decreased appetite (n=278, 123) | 14.7 | 13.0
  New muscle pain (n=324, 151) | 46.9 | 45.0
  Aggravated muscle pain (n=286, 136) | 22.0 | 28.7
  New joint pain (n=278, 128) | 15.5 | 19.5
  Aggravated joint pain (n=272, 131) | 14.0 | 21.4

14. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination 23vPS (Year 0) and 13vPnC / 23vPS (Year 1)
Description: as for outcome 11
Time Frame: as for outcome 6
Population: Safety population; N=number of participants with any systemic event; (n)=number of participants with known values for 23vPS and 13vPnC / 23vPS, respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 23vPS | 13vPnC / 23vPS
Number analyzed (Participants) | 202 | 175
percentage of participants
  Fever: Any ≥38 degrees C (n=127, 129) | 1.6 | 3.1
  Fever: Mild ≥38 but <38.5 degrees C (n=127, 129) | 0.8 | 3.1
  Fever: Moderate ≥38.5 but <39 degrees C(n=127,127) | 0.0 | 0.0
  Fever: Severe ≥39 but ≤40 degrees C(n=127,127) | 0.8 | 0.0
  Fever Potentially life threatening >40C(n=127,127) | 0.0 | 0.0
  Fatigue (n=173, 185) | 49.1 | 51.9
  Headache (n=167, 175) | 46.1 | 49.7
  Chills (n=145, 155) | 26.9 | 29.0
  Rash (n=134, 146) | 13.4 | 24.0
  Vomiting (n=131, 131) | 3.1 | 4.6
  Decreased appetite (n=148, 141) | 23.0 | 17.0
  New muscle pain (n=167, 196) | 51.5 | 61.2
  Aggravated muscle pain (n=154, 164) | 32.5 | 41.5
  New joint pain (n=147, 153) | 23.8 | 25.5
  Aggravated joint pain (n=142, 143) | 21.1 | 17.5

15. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination 2 (Year 1) 13vPnC / 13vPnC, 13vPnC / 23vPS, and 23vPS / 13vPnC
Description: as for outcome 11
Time Frame: 14 days after vaccination 2 (Vax 2=Day 351 up to Day 379 after Visit 1)
Population: Safety population; N=number of participants with any systemic event; (n)=number of participants with known values for 13vPnC / 13vPnC, 13vPnC / 23vPS, and 23vPS / 13vPnC, respectively. Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC / 13vPnC | 13vPnC / 23vPS | 23vPS / 13vPnC
Number analyzed (Participants) | 117 | 222 | 169
percentage of participants
  Fever: Any ≥38 degrees C (n=81, 129, 116) | 2.5 | 3.1 | 0.9
  Fever: Mild ≥38 but <38.5 degrees C (n=81,129,116) | 0.0 | 3.1 | 0.9
  Fever: Moderate ≥38.5, <39 degrees C(n=81,127,115) | 1.2 | 0.0 | 0.0
  Fever: Severe ≥39, ≤40 degrees C(n=81,127,115) | 0.0 | 0.0 | 0.0
  Potentially life threatening >40C(n=81,127,115) | 1.2 | 0.0 | 0.0
  Fatigue (n=100, 185, 141) | 39.0 | 51.9 | 41.1
  Headache (n=96, 175, 139) | 41.7 | 49.7 | 40.3
  Chills (n=90, 155, 127) | 18.9 | 29.0 | 19.7
  Rash (n=86, 146, 121) | 10.5 | 24.0 | 8.3
  Vomiting (n=82, 131, 118) | 3.7 | 4.6 | 6.8
  Decreased appetite (n=89, 141, 123) | 18.0 | 17.0 | 13.0
  New muscle pain (n=108, 196, 151) | 50.0 | 61.2 | 45.0
  Aggravated muscle pain (n=94, 164, 136) | 26.6 | 41.5 | 28.7
  New joint pain (n=87, 153, 128) | 14.9 | 25.5 | 19.5
  Aggravated joint pain (n=91, 143, 131) | 17.6 | 17.5 | 21.4

ADVERSE EVENTS:
Time Frame: Informed consent through 6 Month Follow-up after last vaccination. Local reactions and systemic events assessed within 14 days after vaccination 1 (Vax 1=Day 1/Year 0 [Visit 1]) and 14 days after vaccination 2 (Vax 2=Day 351 up to Day 379 after Visit 1).
Description: Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may=serious for 1 subject and=non-serious for another subject or subject may have experienced both a serious and non-serious episode of same event. AEs/SAEs=non-systematic assessment; local reactions and systemic events=systematic assessment.
Groups:
- 13vPnC (Year 0): Group 1.1: 13vPnC administered as a single dose 0.5 mL IM at Year 0. 13vPnC administered as a single dose 0.5 mL IM at Year 1; or Group 1.2: 13vPnC administered as a single dose 0.5 mL IM at Year 0. 23vPS administered as a single dose 0.5 mL IM at Year 1.
  Other Adverse Events (non-serious events): the number affected (N) for non-systematic (unsolicited) Other Adverse Events N=90; systematic (solicited) Local Reactions N=256; systematic (solicited) Systemic Events N=163.
- 23vPS (Year 0): Group 2: 23vPS administered as a single dose 0.5 mL IM at Year 0. 13vPnC administered as a single dose 0.5 mL IM at Year 1.
  Other Adverse Events (non-serious events): the number affected (N) for non-systematic (unsolicited) Other Adverse Events N=49; systematic (solicited) Local Reactions N=102; systematic (solicited) Systemic Events N=86.
- 13vPnC: 6 Month Follow-up After Vax 1 (Year 0): Group 1.1: 13vPnC administered as a single dose 0.5 mL IM at Year 0. 13vPnC administered as a single dose 0.5 mL IM at Year 1; or Group 1.2: 13vPnC administered as a single dose 0.5 mL IM at Year 0. 23vPS administered as a single dose 0.5 mL IM at Year 1.
- 23vPS: 6 Month Follow-up After Vax 1 (Year 0): Group 2: 23vPS administered as a single dose 0.5 mL IM at Year 0. 13vPnC administered as a single dose 0.5 mL IM at Year 1.
- 13vPnC / 13vPnC (Year 1): 13vPnC administered as a single dose 0.5 mL IM at Year 0. 13vPnC administered as a single dose 0.5 mL IM at Year 1.
  Other Adverse Events (non-serious events): the number affected (N) for non-systematic (unsolicited) Other Adverse Events N=22; systematic (solicited) Local Reactions N=97; systematic (solicited) Systemic Events N=54.
- 13vPnC / 23vPS (Year 1): 13vPnC administered as a single dose 0.5 mL IM at Year 0. 23vPS administered as a single dose 0.5 mL IM at Year 1.
  Other Adverse Events (non-serious events): the number affected (N) for non-systematic (unsolicited) Other Adverse Events N=50; systematic (solicited) Local Reactions N=198; systematic (solicited) Systemic Events N=120.
- 23vPS / 13vPnC (Year 1): 23vPS administered as a single dose 0.5 mL IM at Year 0. 13vPnC administered as a single dose 0.5 mL IM at Year 1.
  Other Adverse Events (non-serious events): the number affected (N) for non-systematic (unsolicited) Other Adverse Events N=32; systematic (solicited) Local Reactions N=118; systematic (solicited) Systemic Events N=68.
- 13vPnC / 13vPnC: 6 Month Follow-up After Vax 2 (Year 1): 13vPnC administered as a single dose 0.5 mL IM at Year 0. 13vPnC administered as a single dose 0.5 mL IM at Year 1.
- 13vPnC / 23vPS: 6 Month Follow-up After Vax 2 (Year 1): 13vPnC administered as a single dose 0.5 mL IM at Year 0. 23vPS administered as a single dose 0.5 mL IM at Year 1.
- 23vPS / 13vPnC: 6 Month Follow-up After Vax 2 (Year 1): 23vPS administered as a single dose 0.5 mL IM at Year 0. 13vPnC administered as a single dose 0.5 mL IM at Year 1.
Arm/Group | 13vPnC (Year 0) | 23vPS (Year 0) | 13vPnC: 6 Month Follow-up After Vax 1 (Year 0) | 23vPS: 6 Month Follow-up After Vax 1 (Year 0) | 13vPnC / 13vPnC (Year 1) | 13vPnC / 23vPS (Year 1) | 23vPS / 13vPnC (Year 1) | 13vPnC / 13vPnC: 6 Month Follow-up After Vax 2 (Year 1) | 13vPnC / 23vPS: 6 Month Follow-up After Vax 2 (Year 1) | 23vPS / 13vPnC: 6 Month Follow-up After Vax 2 (Year 1)
Serious Adverse Events (participants affected / at risk) | 2/478 | 1/237 | 15/478 | 6/237 | 0/160 | 2/267 | 1/223 | 5/160 | 6/267 | 3/223
Other Adverse Events (participants affected / at risk) | 256/478 | 102/237 | 41/478 | 24/237 | 97/160 | 198/267 | 118/223 | 16/160 | 23/267 | 16/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC (Year 0) (N=478) | 23vPS (Year 0) (N=237) | 13vPnC: 6 Month Follow-up After Vax 1 (Year 0) (N=478) | 23vPS: 6 Month Follow-up After Vax 1 (Year 0) (N=237) | 13vPnC / 13vPnC (Year 1) (N=160) | 13vPnC / 23vPS (Year 1) (N=267) | 23vPS / 13vPnC (Year 1) (N=223) | 13vPnC / 13vPnC: 6 Month Follow-up After Vax 2 (Year 1) (N=160) | 13vPnC / 23vPS: 6 Month Follow-up After Vax 2 (Year 1) (N=267) | 23vPS / 13vPnC: 6 Month Follow-up After Vax 2 (Year 1) (N=223)
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis orbital (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian adhesion (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC (Year 0) (N=478) | 23vPS (Year 0) (N=237) | 13vPnC: 6 Month Follow-up After Vax 1 (Year 0) (N=478) | 23vPS: 6 Month Follow-up After Vax 1 (Year 0) (N=237) | 13vPnC / 13vPnC (Year 1) (N=160) | 13vPnC / 23vPS (Year 1) (N=267) | 23vPS / 13vPnC (Year 1) (N=223) | 13vPnC / 13vPnC: 6 Month Follow-up After Vax 2 (Year 1) (N=160) | 13vPnC / 23vPS: 6 Month Follow-up After Vax 2 (Year 1) (N=267) | 23vPS / 13vPnC: 6 Month Follow-up After Vax 2 (Year 1) (N=223)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mixed hyperlipidaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Testicular failure (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Androgen deficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Maculopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/22
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Injection site pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Allergy to vaccine (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 9 | 6 | 0 | 1 | 4 | 4 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 8 | 1 | 0 | 2 | 6 | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 7 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 6 | 1 | 0 | 1 | 3 | 3 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 2 | 0 | 0 | 1 | 4 | 3 | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vascular injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 3 | 1 | 0 | 0 | 2 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Bursa disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sleep disorder due to a general medical condition (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder due to general medical condition, insomnia type (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 0 | 2 | 3 | 2 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Xanthoma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Postmenopause (Social circumstances) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 5 | 0 | 0 | 1 | 2 | 0 | 3 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Orthostatic hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous insufficiency (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Venous valve ruptured (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Redness (Any) (Skin and subcutaneous tissue disorders) | 33/270 | 15/134 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Redness (Any) redness present
Redness (Mild) (Skin and subcutaneous tissue disorders) | 22/266 | 13/134 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Redness (Mild) 2.5 to 5.0 cm
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 17/264 | 5/128 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Redness (Moderate) 5.1 to 10.0 cm
Redness (Severe) (Skin and subcutaneous tissue disorders) | 3/259 | 1/127 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Redness (Severe) >10 cm
Swelling (Any) (Skin and subcutaneous tissue disorders) | 27/270 | 14/135 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Swelling (Any) swelling present
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 22/268 | 8/132 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Swelling (Mild) 2.5 to 5.0 cm
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 10/263 | 10/132 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Swelling (Moderate) 5.1 to 10.0 cm
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/258 | 0/127 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Swelling (Severe) >10 cm
Pain (Any) (Skin and subcutaneous tissue disorders) | 256/370 | 102/175 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Pain (Any) pain present
Pain (Mild) (Skin and subcutaneous tissue disorders) | 238/360 | 90/170 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Pain (Mild) awareness of pain; easily tolerated
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 57/284 | 31/143 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Pain (Moderate) discomfort enough to cause interference with usual activity
Pain (Severe) (Skin and subcutaneous tissue disorders) | 6/261 | 1/127 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Pain (Severe) incapacitating
Limitation of arm movement (Any) (Skin and subcutaneous tissue disorders) | 68/289 | 40/142 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Limitation of arm movement (Any) limitation present
Limitation of arm movement (Mild) (Skin and subcutaneous tissue disorders) | 65/286 | 37/142 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Limitation of arm movement (Mild) some limitation
Limitation of arm movement (Moderate) (Skin and subcutaneous tissue disorders) | 3/260 | 4/127 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Limitation of arm movement (Moderate) unable to move arm above head; able to move arm above shoulder
Limitation of arm movement (Severe) (Skin and subcutaneous tissue disorders) | 3/261 | 3/128 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Limitation of arm movement (Severe) unable to move arm above shoulder
Redness (Any) (Skin and subcutaneous tissue disorders) | 9/61 | 0/0 | 0/0 | 0/0 | 7/61 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Redness (Any)
Redness (Mild) (Skin and subcutaneous tissue disorders) | 4/57 | 0/0 | 0/0 | 0/0 | 5/57 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Redness (Mild)
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 5/58 | 0/0 | 0/0 | 0/0 | 2/58 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Redness (Moderate)
Redness (Severe) (Skin and subcutaneous tissue disorders) | 0/57 | 0/0 | 0/0 | 0/0 | 2/57 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Redness (Severe)
Swelling (Any) (Skin and subcutaneous tissue disorders) | 6/60 | 0/0 | 0/0 | 0/0 | 7/60 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Swelling (Any)
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 4/59 | 0/0 | 0/0 | 0/0 | 5/59 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Swelling (Mild)
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 1/55 | 0/0 | 0/0 | 0/0 | 2/55 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Swelling (Moderate)
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/56 | 0/0 | 0/0 | 0/0 | 1/56 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Swelling (Severe)
Pain (Any) (Skin and subcutaneous tissue disorders) | 83/108 | 0/0 | 0/0 | 0/0 | 82/108 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Pain (Any)
Pain (Mild) (Skin and subcutaneous tissue disorders) | 73/101 | 0/0 | 0/0 | 0/0 | 73/101 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Pain (Mild)
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 13/61 | 0/0 | 0/0 | 0/0 | 16/61 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Pain (Moderate)
Pain (Severe) (Skin and subcutaneous tissue disorders) | 0/57 | 0/0 | 0/0 | 0/0 | 2/57 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Pain (Severe)
Limitation of arm movement (Any) (Skin and subcutaneous tissue disorders) | 17/65 | 0/0 | 0/0 | 0/0 | 16/65 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Limitation of arm movement (Any)
Limitation of arm movement (Mild) (Skin and subcutaneous tissue disorders) | 17/65 | 0/0 | 0/0 | 0/0 | 16/65 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Limitation of arm movement (Mild)
Limitation of arm movement (Moderate) (Skin and subcutaneous tissue disorders) | 1/56 | 0/0 | 0/0 | 0/0 | 0/56 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Limitation of arm movement (Moderate)
Limitation of arm movement (Severe) (Skin and subcutaneous tissue disorders) | 0/56 | 0/0 | 0/0 | 0/0 | 1/56 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Limitation of arm movement (Severe)
Redness (Any) (Skin and subcutaneous tissue disorders) | 33/270 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 5/115 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Redness (Any)
Redness (Mild) (Skin and subcutaneous tissue disorders) | 22/266 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 5/115 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Redness (Mild)
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 17/264 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1/115 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Redness (Moderate)
Redness (Severe) (Skin and subcutaneous tissue disorders) | 3/259 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/115 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Redness (Severe)
Swelling (Any) (Skin and subcutaneous tissue disorders) | 27/270 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 6/119 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Swelling (Any)
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 22/268 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 6/119 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Swelling (Mild)
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 10/263 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1/116 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Swelling (Moderate)
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/258 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/115 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Swelling (Severe)
Pain (Any) (Skin and subcutaneous tissue disorders) | 256/370 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 118/169 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Pain (Any)
Pain (Mild) (Skin and subcutaneous tissue disorders) | 238/360 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 113/166 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Pain (Mild)
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 57/284 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 23/129 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Pain (Moderate)
Pain (Severe) (Skin and subcutaneous tissue disorders) | 6/261 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1/116 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Pain (Severe)
Limitation of arm movement (Any) (Skin and subcutaneous tissue disorders) | 68/289 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 24/130 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Limitation of arm movement (Any)
Limitation of arm movement (Mild) (Skin and subcutaneous tissue disorders) | 65/286 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 22/130 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Limitation of arm movement (Mild)
Limitation of arm movement (Moderate) (Skin and subcutaneous tissue disorders) | 3/260 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/115 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Limitation of arm movement (Moderate)
Limitation of arm movement (Severe) (Skin and subcutaneous tissue disorders) | 3/261 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 2/115 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Limitation of arm movement (Severe)
Redness (Any) (Skin and subcutaneous tissue disorders) | 0/0 | 15/134 | 0/0 | 0/0 | 0/0 | 42/151 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Redness (Any)
Redness (Mild) (Skin and subcutaneous tissue disorders) | 0/0 | 13/134 | 0/0 | 0/0 | 0/0 | 28/144 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Redness (Mild)
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 0/0 | 5/128 | 0/0 | 0/0 | 0/0 | 17/138 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Redness (Moderate)
Redness (Severe) (Skin and subcutaneous tissue disorders) | 0/0 | 1/127 | 0/0 | 0/0 | 0/0 | 9/131 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Redness (Severe)
Swelling (Any) (Skin and subcutaneous tissue disorders) | 0/0 | 14/135 | 0/0 | 0/0 | 0/0 | 40/155 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Swelling (Any)
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 0/0 | 8/132 | 0/0 | 0/0 | 0/0 | 30/149 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Swelling (Mild)
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 0/0 | 10/132 | 0/0 | 0/0 | 0/0 | 17/138 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Swelling (Moderate)
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/0 | 0/127 | 0/0 | 0/0 | 0/0 | 8/132 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Swelling (Severe)
Pain (Any) (Skin and subcutaneous tissue disorders) | 0/0 | 102/175 | 0/0 | 0/0 | 0/0 | 198/231 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Pain (Any)
Pain (Mild) (Skin and subcutaneous tissue disorders) | 0/0 | 90/170 | 0/0 | 0/0 | 0/0 | 161/205 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Pain (Mild)
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 0/0 | 31/143 | 0/0 | 0/0 | 0/0 | 87/176 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Pain (Moderate)
Pain (Severe) (Skin and subcutaneous tissue disorders) | 0/0 | 1/127 | 0/0 | 0/0 | 0/0 | 18/140 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Pain (Severe)
Limitation of arm movement (Any) (Skin and subcutaneous tissue disorders) | 0/0 | 40/142 | 0/0 | 0/0 | 0/0 | 95/178 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Limitation of arm movement (Any)
Limitation of arm movement (Mild) (Skin and subcutaneous tissue disorders) | 0/0 | 37/142 | 0/0 | 0/0 | 0/0 | 81/171 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Limitation of arm movement (Mild)
Limitation of arm movement (Moderate) (Skin and subcutaneous tissue disorders) | 0/0 | 4/127 | 0/0 | 0/0 | 0/0 | 14/134 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Limitation of arm movement (Moderate)
Limitation of arm movement (Severe) (Skin and subcutaneous tissue disorders) | 0/0 | 3/128 | 0/0 | 0/0 | 0/0 | 11/135 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Limitation of arm movement (Severe)
Redness (Any) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 11/86 | 42/151 | 5/115 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Redness (Any)
Redness (Mild) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 6/83 | 28/144 | 5/115 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Redness (Mild)
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 6/83 | 17/138 | 1/115 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Redness (Moderate)
Redness (Severe) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 2/83 | 9/131 | 0/115 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Redness (Severe)
Swelling (Any) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 12/86 | 40/155 | 6/119 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Swelling (Any)
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 9/85 | 30/149 | 6/119 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Swelling (Mild)
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 5/82 | 17/138 | 1/116 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Swelling (Moderate)
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 1/82 | 8/132 | 0/115 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Swelling (Severe)
Pain (Any) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 97/129 | 198/231 | 118/169 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Pain (Any)
Pain (Mild) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 89/123 | 161/205 | 113/166 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Pain (Mild)
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 22/91 | 87/176 | 23/129 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Pain (Moderate)
Pain (Severe) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 2/83 | 18/140 | 1/116 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Pain (Severe)
Limitation of arm movement (Any) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 26/93 | 95/178 | 24/130 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Limitation of arm movement (Any)
Limitation of arm movement (Mild) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 25/92 | 81/171 | 22/130 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Limitation of arm movement (Mild)
Limitation of arm movement (Moderate) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 3/83 | 14/134 | 0/115 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Limitation of arm movement (Moderate)
Limitation of arm movement (Severe) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 1/82 | 11/135 | 2/115 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Limitation of arm movement (Severe)
Fever (Any) (General disorders) | 12/263 | 2/127 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Fever (Any) ≥38 degrees C
Fever (Mild) (General disorders) | 10/263 | 1/127 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Fever (Mild) ≥38 but <38.5 degrees C
Fever (Moderate) (General disorders) | 2/259 | 0/127 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Fever (Moderate) ≥38.5 but <39 degrees C
Fever (Severe) (General disorders) | 1/259 | 1/127 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Fever (Severe) ≥39 but ≤40 degrees C
Fever (Potentially life threatening) (General disorders) | 1/258 | 0/127 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Fever (Potentially life threatening) >40C
Fatigue (General disorders) | 162/321 | 85/173 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Fatigue
Headache (General disorders) | 163/328 | 77/167 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Headache
Chills (General disorders) | 57/286 | 39/145 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Chills
Rash (General disorders) | 23/267 | 18/134 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Rash
Vomiting (General disorders) | 8/261 | 4/131 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Vomiting
Decreased appetite (General disorders) | 41/278 | 34/148 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Decreased appetite
New generalized muscle pain (General disorders) | 152/324 | 86/167 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; New generalized muscle pain
Aggravated generalized muscle pain (General disorders) | 63/286 | 50/154 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Aggravated generalized muscle pain
New generalized joint pain (General disorders) | 43/278 | 35/147 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; New generalized joint pain
Aggravated generalized joint pain (General disorders) | 38/272 | 30/142 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC and 23vPS Year 0; Aggravated generalized joint pain
Fever (Any) (General disorders) | 5/55 | 0/0 | 0/0 | 0/0 | 2/55 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Fever (Any)
Fever (Mild) (General disorders) | 4/55 | 0/0 | 0/0 | 0/0 | 0/55 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Fever (Mild)
Fever (Moderate) (General disorders) | 0/55 | 0/0 | 0/0 | 0/0 | 1/55 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Fever (Moderate)
Fever (Severe) (General disorders) | 0/55 | 0/0 | 0/0 | 0/0 | 0/55 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Fever (Severe)
Fever (Potentially life threatening) (General disorders) | 1/55 | 0/0 | 0/0 | 0/0 | 1/55 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Fever (Potentially life threatening)
Fatigue (General disorders) | 43/76 | 0/0 | 0/0 | 0/0 | 33/76 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Fatigue
Headache (General disorders) | 40/76 | 0/0 | 0/0 | 0/0 | 34/76 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Headache
Chills (General disorders) | 11/61 | 0/0 | 0/0 | 0/0 | 12/61 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Chills
Rash (General disorders) | 5/60 | 0/0 | 0/0 | 0/0 | 6/60 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Rash
Vomiting (General disorders) | 4/56 | 0/0 | 0/0 | 0/0 | 2/56 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Vomiting
Decreased appetite (General disorders) | 8/61 | 0/0 | 0/0 | 0/0 | 13/61 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Decreased appetite
New generalized muscle pain (General disorders) | 40/84 | 0/0 | 0/0 | 0/0 | 43/84 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); New generalized muscle pain
Aggravated generalized muscle pain (General disorders) | 18/68 | 0/0 | 0/0 | 0/0 | 21/68 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Aggravated generalized muscle pain
New generalized joint pain (General disorders) | 9/62 | 0/0 | 0/0 | 0/0 | 10/62 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); New generalized joint pain
Aggravated generalized joint pain (General disorders) | 10/62 | 0/0 | 0/0 | 0/0 | 12/62 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 13vPnC / 13vPnC (Year 1); Aggravated generalized joint pain
Fever (Any) (General disorders) | 12/263 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1/116 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Fever (Any)
Fever (Mild) (General disorders) | 10/263 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1/116 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Fever (Mild)
Fever (Moderate) (General disorders) | 2/259 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/115 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Fever (Moderate)
Fever (Severe) (General disorders) | 1/259 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/115 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Fever (Severe)
Fever (Potentially life threatening) (General disorders) | 1/258 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/115 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Fever (Potentially life threatening)
Fatigue (General disorders) | 162/321 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 58/141 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Fatigue
Headache (General disorders) | 163/328 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 56/139 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Headache
Chills (General disorders) | 57/286 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 25/127 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Chills
Rash (General disorders) | 23/267 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 10/121 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Rash
Vomiting (General disorders) | 8/261 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 8/118 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Vomiting
Decreased appetite (General disorders) | 41/278 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 16/123 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Decreased appetite
New generalized muscle pain (General disorders) | 152/324 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 68/151 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); New generalized muscle pain
Aggravated generalized muscle pain (General disorders) | 63/286 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 39/136 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Aggravated generalized muscle pain
New generalized joint pain (General disorders) | 43/278 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 25/128 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); New generalized joint pain
Aggravated generalized joint pain (General disorders) | 38/272 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 28/131 | 0/0 | 0/0 | 0/0 — 13vPnC (Year 0) and 23vPS / 13vPnC (Year 1); Aggravated generalized joint pain
Fever (Any) (General disorders) | 0/0 | 2/127 | 0/0 | 0/0 | 0/0 | 4/129 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Fever (Any)
Fever (Mild) (General disorders) | 0/0 | 1/127 | 0/0 | 0/0 | 0/0 | 4/129 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Fever (Mild)
Fever (Moderate) (General disorders) | 0/0 | 0/127 | 0/0 | 0/0 | 0/0 | 0/127 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Fever (Moderate)
Fever (Severe) (General disorders) | 0/0 | 1/127 | 0/0 | 0/0 | 0/0 | 0/127 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Fever (Severe)
Fever (Potentially life threatening) (General disorders) | 0/0 | 0/127 | 0/0 | 0/0 | 0/0 | 0/127 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Fever (Potentially life threatening)
Fatigue (General disorders) | 0/0 | 85/173 | 0/0 | 0/0 | 0/0 | 96/185 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Fatigue
Headache (General disorders) | 0/0 | 77/167 | 0/0 | 0/0 | 0/0 | 87/175 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Headache
Chills (General disorders) | 0/0 | 39/145 | 0/0 | 0/0 | 0/0 | 45/155 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Chills
Rash (General disorders) | 0/0 | 18/134 | 0/0 | 0/0 | 0/0 | 35/146 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Rash
Vomiting (General disorders) | 0/0 | 4/131 | 0/0 | 0/0 | 0/0 | 6/131 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Vomiting
Decreased appetite (General disorders) | 0/0 | 34/148 | 0/0 | 0/0 | 0/0 | 24/141 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Decreased appetite
New generalized muscle pain (General disorders) | 0/0 | 86/167 | 0/0 | 0/0 | 0/0 | 120/196 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); New generalized muscle pain
Aggravated generalized muscle pain (General disorders) | 0/0 | 50/154 | 0/0 | 0/0 | 0/0 | 68/164 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Aggravated generalized muscle pain
New generalized joint pain (General disorders) | 0/0 | 35/147 | 0/0 | 0/0 | 0/0 | 39/153 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); New generalized joint pain
Aggravated generalized joint pain (General disorders) | 0/0 | 30/142 | 0/0 | 0/0 | 0/0 | 25/143 | 0/0 | 0/0 | 0/0 | 0/0 — 23vPS (Year 0) and 13vPnC / 23vPS (Year 1); Aggravated generalized joint pain
Fever (Any) (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 2/81 | 4/129 | 1/116 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Fever (Any)
Fever (Mild) (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/81 | 4/129 | 1/116 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Fever (Mild)
Fever (Moderate) (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 1/81 | 0/127 | 0/115 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Fever (Moderate)
Fever (Severe) (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/81 | 0/127 | 0/115 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Fever (Severe)
Fever (Potentially life threatening) (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 1/81 | 0/127 | 0/115 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Fever (Potentially life threatening)
Fatigue (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 39/100 | 96/185 | 58/141 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Fatigue
Headache (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 40/96 | 87/175 | 56/139 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Headache
Chills (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 17/90 | 45/155 | 25/127 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Chills
Rash (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 9/86 | 35/146 | 10/121 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Rash
Vomiting (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 3/82 | 6/131 | 8/118 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Vomiting
Decreased appetite (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 16/89 | 24/141 | 16/123 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Decreased appetite
New generalized muscle pain (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 54/108 | 120/196 | 68/151 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); New generalized muscle pain
Aggravated generalized muscle pain (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 25/94 | 68/164 | 39/136 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Aggravated generalized muscle pain
New generalized joint pain (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 13/87 | 39/153 | 25/128 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); New generalized joint pain
Aggravated generalized joint pain (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 16/91 | 25/143 | 28/131 | 0/0 | 0/0 | 0/0 — 13vPnC / 13vPnC (Year 1), 13vPnC / 23vPS (Year 1), and 23vPS / 13vPnC (Year 1); Aggravated generalized joint pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.